CLINICAL TRIAL: NCT01364857
Title: French National Prospective Cohort of Children With Port Wine Stain on a Limb = "Cohorte Nationale d'Enfants Avec Angiome Plan de Membre inférieur"
Brief Title: French National Cohort of Children With Port Wine Stain
Acronym: CONAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PHRN09 - GL / CONAPE
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2023-08

CONDITIONS: Port Wine Stain; Klippel Trenaunay Syndrome; Parkes Weber Syndrome
Keywords: port wine stain of a limb
MeSH Terms: conditions — Port-Wine Stain; Klippel-Trenaunay-Weber Syndrome; Sturge-Weber Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PWS cohort (Other): search for polymorphisms of RASA1 gene
  Interventions: Genetic: search for polymorphisms of RASA1 gene

INTERVENTIONS:
Genetic: search for polymorphisms of RASA1 gene — Blood sample ( 5 mL) at tne inclusion of the child DNA extraction and genetic analysis of the 24 exons of RASA1 gene after specific consent

SUMMARY:
Port Wine Stain on a limb can be either isolated or associated with complications (venous or orthopedic impairment, arteriovenous malformations), leading sometimes to complex syndromes (Klippel-Trenaunay syndrome,Parkes-Weber syndrome).

Little is known about epidemiology of port wine stains: their evolution during the growth of the child, the frequency of complications, genetic data, and prognostic factors.

This prospective french national cohort will help for : description of the evolution of port wine stain and possible complications; prognostic factors for complications ; association with mutations of RASA1 gene; quality of life of these children. It will also help for global appreciation of the management of this disease in France.

DETAILED DESCRIPTION:
Prospective national study, including 16 Pediatric and Dermatologic Departments.

Methods : each children with a port wine stain on a lower limb will be followed up for 5 years.

Collected data : demographic data, clinical features, alterations of RASA1 gene, vascular evaluation by ultrasonographic and orthopedic evaluation by X rays, quality of life with a questionnaire.

Inclusion period = 3 years Follow up period = 5 years Population = 150 children

ELIGIBILITY:
Inclusion Criteria:

* Child between 2 and 12 years old with a port wine stain on a lower limb ( or two lower limbs) with national health assurance with consent from one parent

Exclusion Criteria:

* child with orthopedic impairment with no link with the port wine stain

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Complicated evolution (defined as: vascular, orthopedic or systemic involvement linked with the port wine stain) | during the 5 years of follow up
  Complicated evolution (defined as: vascular, orthopedic or systemic involvement linked with the port wine stain)

SECONDARY OUTCOMES:
Mutations of RASA 1 gene | during the 5 years of follow up
  Mutations of RASA 1 gene

CONTACTS AND LOCATIONS:
Overall Officials: Violaine MIZZI, Study Chair — University Hospital, Tours
Locations (17):
- France (17):
  - Service de dermatologie, Amiens
  - Service de dermatologie, Angers
  - Service de dermatologie, Bordeaux
  - Service de dermatologie, Caen
  - Service de dermatologie, Dijon
  - Service de Dermatologie, Bâtiment tardieu, Le Mans
  - Service de Dermatologie, Hôpital St Eloi, Montpellier
  - Service de dermatologie, Nantes
  - Service de dermatologie, Nice
  - Service de dermatologie, Paris
  - Service de dermatlogie, Quimper
  - Service de dermatologie, Reims
  - Service de Dermatologie, Hôpital Pontchaillou, CHU de Rennes, Rennes
  - Service de dermatologie, Rouen
  - Service de dermatologie, Saint-Etienne
  - Service de dermatologie, Toulouse
  - Service de dermatologie, Tours

REFERENCES:
- [Result] Maruani A, Durieux-Verde M, Mazereeuw-Hautier J, Boccara O, Martin L, Chiaverini C, Eschard C, Beneton N, Vabres P, Balguerie X, Plantin P, Bessis D, Barbarot S, Dadban A, Droitcourt C, Berthelot A, Lorette G, Leducq S, Samimi M, Andres C, Caille A, Vourc'h P; Groupe de Recherche de la Societe Francaise de Dermatologie. Search for RASA1 Variants in Capillary Malformations of the Legs in 113 Children: Results from the French National Paediatric Cohort CONAPE. Acta Derm Venereol. 2018 Feb 7;98(2):251-255. doi: 10.2340/00015555-2835. PMID 29110021